CLINICAL TRIAL: NCT00003663
Title: Rituximab Anti-CD20 Monoclonal Antibody and Dexamethasone in the Treatment of Relapsed Indolent Lymphoma
Brief Title: Rituximab and Dexamethasone in Treating Patients With Recurrent or Refractory Indolent Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no patient accrual
Sponsor: Hoag Memorial Hospital Presbyterian (Other)
Collaborators: Cancer Biotherapy Research Group (Other)
Responsible Party: Robert O. Dillman, MD, Hoag Memorial Hospital Presbyterian
Purpose: Treatment
Other Study IDs: CDR0000066756; CBRG-9805; NCI-V98-1492
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Lymphoma
Keywords: Waldenstrom macroglobulinemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Waldenstrom Macroglobulinemia; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: rituximab
Drug: dexamethasone

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining the monoclonal antibody rituximab with dexamethasone may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of rituximab and dexamethasone in treating patients with recurrent or refractory indolent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxic effects of rituximab and dexamethasone in patients with recurrent or refractory indolent non-Hodgkin's lymphoma. II. Determine the objective tumor response rate and duration of response at 2 months after initiation of therapy, and the percentage of patients with progressive disease. III. Determine the maximum response, duration of response, and progression free interval for patients who have not progressed after 4 weeks of therapy. IV. Determine the failure-free and overall survival of these patients on this regimen. V. Compare the response rate and survival rates to results for similar patients (historical and concurrent) who have received 4 weeks of rituximab without dexamethasone, and patients who did not receive maintenance rituximab.

OUTLINE: Patients receive dexamethasone IV followed by rituximab IV on days 1, 8, 15, and 22 for one course. Two months after initiating treatment, patients are evaluated for disease progression. Patients with stable or responding disease may receive monthly dexamethasone and rituximab therapy for up to 10 additional months. Patients are followed every 3 months for 2 years, then every 6 months for years 3-4, and then yearly for up to 5 years.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven stage III or IV, recurrent or refractory, indolent B cell non-Hodgkin's lymphoma of the following types: Working Group Formulation A (small cell lymphocytic) Working Group Formulation B, C, and D (follicular) Must have relapsed after prior chemotherapy At least 1 lymph node or visceral lesion at least 2 cm in diameter

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: Lymphocyte count less than 5,000/mm3 Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Fertile patients must use effective contraception No active infection HIV negative No hepatitis B or C No concurrent life threatening condition

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior monoclonal antibody therapy for lymphoma (e.g., rituximab) Chemotherapy: See Disease Characteristics Endocrine therapy: No other concurrent corticosteroids and/or epinephrine (unless anaphylactic shock) Radiotherapy: Not specified Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 1998-06; Primary Completion 2000-01 (Actual); Study Completion 2000-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Study Chair — Cancer Biotherapy Research Group
Locations (3):
- United States (3):
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - Cancer Care Center for Southern Indiana, Bloomington, Indiana
  - St. Joseph Regional Cancer Center, Bryan, Texas